CLINICAL TRIAL: NCT00588471
Title: The Effect of Acute Statin Treatment on Inflammation and Peripheral Arterial Tone in Patients Undergoing Percutaneous Coronary Intervention.
Brief Title: Effect of Acute Statin Treatment in Patients Undergoing Percutaneous Coronary Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because not enough subjects could be recruited.
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Amir Lerman, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2026-02
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Active Comparator): Subjects randomized to this arm will be pretreated with 80 mg (2 pills) simvastatin approximately one hour prior to percutaneous coronary intervention.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Subjects randomized to this arm will be pretreated with 2 placebo pills approximately one hour prior to percutaneous coronary intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Subjects randomized to this arm will be pretreated with 80 mg (2 pills) simvastatin approximately one hour prior to percutaneous coronary intervention.
  Other Names: Zocar
  Arms: Simvastatin
Drug: Placebo — Subjects randomized to this arm will be pretreated with 2 placebo pills approximately one hour prior to percutaneous coronary intervention.
  Arms: Placebo

SUMMARY:
The goal of this study is to determine if one dose of simvastatin will decrease the inflammatory response to coronary intervention. Also to determine if one dose of simvastatin affects endothelial function (activity of the artery) as measured by noninvasive peripheral artery tonography.

DETAILED DESCRIPTION:
The objective of this study is to determine if acute pretreatment with simvastatin, an HMG-CoA reductase inhibitor will reduce the post inflammatory response after percutaneous coronary interventions (PCI), and/or change endothelial function as assessed by peripheral arterial tomography (PAT). Percutaneous coronary intervention (PCI), commonly known as coronary angioplasty or simply angioplasty, is a non-surgical procedure used to treat the stenotic (narrowed) coronary arteries of the heart found in coronary heart disease.

Patients will be pretreated with simvastatin 80 mg prior to undergoing PCI. Endothelial function will be assessed before and after treatment via PAT. Our working hypothesis is patients pretreated with simvastatin, will have 1) attenuated inflammatory response, as noted by decreased levels of serum high sensitivity CRP and IL-6 and 2) improved endothelial function as compared to patients not pretreated with statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PCI/angiography
* No previously known side effects of statins
* Patients who sign an informed consent
* Age > 18 years old

Exclusion Criteria:

* Patients with ST elevation myocardial infarction
* Patients with cardiogenic shock
* Patients with hypersensitivity to statins
* Patients with unexplained muscle pain
* Patients with acute liver disease
* Patients receiving cyclosporine, antifungal azoles, macrolide antibiotics, niacin, fibrates> 1 quart grapefruit juice/day or nefazodone
* Patients with creatinine > 2.0
* Patients with known malignancy
* Ejection Fraction < 25%
* No coronary care unit patients
* No outpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at the Mayo Clinic in Rochester, MN from 2002 until 2008.
Pre-assignment Details: 66 subjects signed informed consent, but 9 subjects had to have the PCI procedure too quickly, and could not participate in the study.
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 28 | 29
Completed | 28 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 11 | 15 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum High Sensitivity C-Reactive Protein (hsCRP)
Description: The hsCRP test evaluates vascular inflammation. People with higher hsCRP values have the highest risk of cardiovascular disease, and those with lower values have less of a risk. The American Heart Association and U.S. Centers for Disease Control and Prevention have defined risk groups as follows:
  Low risk: less than 1.0 mg/L Average risk: 1.0 to 3.0 mg/L High risk: above 3.0 mg/L
Time Frame: baseline, within 24 hours post percutaneous coronary intervention
Population: The study was terminated early because not enough subjects could be recruited.
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Endothelial Peripheral Arterial Tomography (EndoPAT) Score After PCI
Description: The EndoPAT is a noninvasive test that involves putting probes on the index fingers of both hands and evaluating the blood flow to one hand before and after inflating a blood pressure cuff on one arm, temporarily reducing blood flow to the fingers. The finger sensor on the affected arm will now show no blood flow, while the sensor on the opposite index finger will continue to display your normal blood flow level. After several minutes, the blood pressure cuff is released, allowing blood to flow back into the affected lower arm. If the finger sensor on the affected arm shows a rush of blood, the blood vessels are functioning normally. If the blood flow return is sluggish, however, the blood vessels are unhealthy.
  The results are reported as the "Endoscore" (range 0-3); a score of 1.67 and lower indicates the need for immediate medical attention; a score between 1.68 and 2 indicates a need to reduce risk factors; a score above 2.1 indicates a healthy heart.
Time Frame: baseline, within 24 hours post percutaneous coronary intervention
Population: The study was terminated early because not enough subjects could be recruited.
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events will be carefully monitored while the subject is on the study medicine, within 24 hours after the coronary procedure.
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 1/28 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=28) | Placebo (N=29)
Subject could not tolerate the Blood Pressure Cuff (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early because not enough subjects could be recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No